CLINICAL TRIAL: NCT02454803
Title: An International, Multicentre, Observational, Prospective, Longitudinal Cohort Study to Assess the Impact of Integrated Upper Limb Spasticity Management Including the Use of BoNT-A- Injections on Patient-centred Goal Attainment in Real Life Practice - ULIS III
Brief Title: Attainment of Person-centred Goals After Botulinum Toxin Treatment for Upper Limb Spasticity in Real Life Practice
Acronym: ULIS III
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: Y-79-52120-206
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Upper Limb Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose for this study is to understand the effect of botulinum toxin as a treatment integrated in the management of spasticity (stiffness) in the arm and/or hand, arising from any neurological condition. The study will look at the types of goals that people choose for treatment, and the extent to which these are achieved in different individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with ULS, in whom a decision has already been made to inject botulinum toxin A (BoNT A).
* Patient has provided written informed consent for collection of the data.

Exclusion Criteria:

* Participation in any interventional clinical study of ULS within the 12 weeks prior to the inclusion visit (Visit 1).
* Patient has already been included in the current study, but was subsequently withdrawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient suffering from upper limb spasticity (ULS) seen in clinic, hospital and/or rehabilitation centers.
Sampling Method: Non-Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2015-01; Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Patient centred goal attainment will be assessed using the cumulated Goal Attainment Scale Total Score (GAS T score). | From visit 1 (injection 1) and up to the end of the study (maximum 24 months after first injection)
  Goal attainment will be recorded on a five point numerical scale (range -2 to +2) and goal scores combined to give an aggregated T score.

SECONDARY OUTCOMES:
To document the baseline patient characteristics and disease history. | Baseline
  Muscle tone will be evaluated using the Modified Ashworth Scale (MAS). Severity of different aspects of impairment in patients with neurological damage will be evaluated using the Upper Limb Spasticity Neurological Impairment Scale (ULS-NIS) recorded for both upper limbs.
To document the clinical management of the upper limb spasticity. | From visit 1 (injection 1) and up to the end of the study (maximum 24 months after first injection)
  BoNT-A injection practices, concomitant drug and non-drug therapies.
Patient centred goal attainment by goal area. | From visit 1 (injection 1) and up to the end of the study (maximum 24 months after first injection)
  Assessed using the cumulated GAS T score of all goals assessed within each goal area.
Evolution of goal changes across the study will be recorded alongside changes from baseline in the standardised outcome measures. | From visit 1 (injection 1) and up to the end of the study (maximum 24 months after first injection)
Assessment of the correlations between patient centred goals and related standardised rating scales. | From visit 1 (injection 1) and up to the end of the study (maximum 24 months after first injection)
  Using Goal Attainment Scaling Evaluation of Intensity (GASeous) and standardised outcome measures.
Evaluation of change from baseline in the four domains of Disability Assessment Scale (DAS) as well as in the Principal Target of Treatment (PTT). | From visit 1 (injection 1) and up to the end of the study (maximum 24 months after first injection)
  The DAS will be used at each visit to determine the extent of functional impairment in four domains: hygiene, dressing, limb position and pain. Impairment is assessed on a four point scale (range 0 to 3, where 0=no disability, and 3=severe disability). The PTT will be defined at each visit, based on one of the four DAS domains.
Evolution of quality of life | From visit 1 (injection 1) and up to the end of the study (maximum 24 months after first injection)
  Assessed at each visit in a subpopulation of English-native speaker patients in Anglophone countries based on two different quality of life instruments, EuroQol 5 Dimensions, 5 levels (EQ 5D 5L) and Spasticity Related Quality of Life Tool (SQoL 6D).
Health economic | From visit 1 (injection 1) and up to the end of the study (maximum 24 months after first injection)
  Health economic analysis will include changes in concomitant treatments, changes in patient employment status, maintenance of health care (by nurse, caregiver etc) and utility data derived from EQ-5D 5L, DAS, GAS and SQoL-6D.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (57):
- United States (5):
  - Design Neuroscience, Doral, Florida
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Kansas City Bone & Joint Clinic, Overland Park, Kansas
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Vanderbilt University, Nashville, Tennessee
- Australia (9):
  - Epworth Rehabilitation Camberwell, Camberwell
  - St Vincent's Hospital, Darlinghurst
  - Austin Health Hospital, Heidelberg
  - Liverpool Brain Injury Rehabilitation Unit, Liverpool
  - Royal Melbourne Hospital, Parkville
  - Prince of Wales Hospital, Randwick
  - RPAH, Sydney
  - Westmead Hospital, Westmead
  - Princess Alexandra Hospital, Woolloongabba
- Gaitlal-Klinik Hermagor, Hermagor, Austria
- Brazil (3):
  - Hospital de Clinicas da UFPR, Curitiba
  - Fundacao Faculdade Regional de Medicina, São José do Rio Preto
  - Hospital dos Clinicas Universitaria de Sao Paulo, São Paulo
- France (5):
  - Centre Régional de Rééducation et Réadaptation Fonctionnelle, Angers
  - CHU Pellegrin, Bordeaux
  - Hôpital Raymond Poincaré, Garches
  - CHU Grenoble Hôpital Sud, Grenoble
  - Institut Universitaire de Réadaptation de Clémenceau, Strasbourg
- Germany (5):
  - Universitaets-Klinikum Erlangen, Erlangen
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum rechts der Isar der Technischen Universitaet Muenchen, Munich
  - Schoen Klinik Muenchen Schwabing, Munich
  - Universitaetsklinikum Wuerzburg, Würzburg
- Tung Wah Hospital, Hong Kong, Hong Kong
- Italy (7):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari
  - Ospedale Valduce - Villa Beretta, Costa Masnaga
  - Azienda Ospedaliero Universitaria di Ferrara, Ferrara
  - Azienda Ospedaliero Universitaria Policlinico "G Martino", Messina
  - Fondazione Santa Lucia, I.R.C.C.S., Roma
  - Fondazione Don Carlo Gnocchi Onlus, Sarzana
- Mexico (4):
  - Hospital Angeles Clinica Londres, Mexico City
  - Grupo Torre Medica, México
  - National Institute of Neurology/Rehabilitation, México
  - Rehabilitation Centre, Querétaro
- Philippines (2):
  - Perpetual Succour Hospital, Cebu City
  - Metropolitan Medical Center, Manila
- Poland (3):
  - Academy of Neurology, Krakow
  - Bonacha, Warsaw
  - Public Hospital Wojewodzki, Warsaw
- Portugal (3):
  - Alcoitao Rehabilitation Centre, Alcoitão
  - Hospital de Faro, Faro
  - Hospital Egas Moniz, Lisbon
- Russia (7):
  - Regional State Budgetary Healthcare Institution "City Hospital N°5", Barnaul
  - Interregional Cinical and Diagnostic Centre, Kazan'
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - Krasnoyarsks State Medical University, Krasnoyarsk
  - Federal State Hospital for Treatment and Rehabilitation, Moscow
  - Federal State Budgetary Institution, Saint Petersburg
  - Pavlov First Saint-Petersburg State Medical University, Saint Petersburg
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - Veteran General Hospital, Taipei

REFERENCES:
- [Derived] Khat'kova SE, Baikova A, Maisonobe P, Khasanova DR. [Impact of integrated upper limb spasticity management including repeat botulinum toxin type A (BoNT-A) injections on patient-centred goal attainment in real-life practice: results from the prospective, observational Upper Limb International Spasticity cohort study (ULIS-III) in a Russian subpopulation]. Zh Nevrol Psikhiatr Im S S Korsakova. 2021;121(11):39-48. doi: 10.17116/jnevro202112111139. Russian. PMID 34932284
- [Derived] Turner-Stokes L, Jacinto J, Fheodoroff K, Brashear A, Maisonobe P, Lysandropoulos A, Ashford S; Upper Limb International Spasticity-III (ULIS-III) study group. Assessing the effectiveness of upper-limb spasticity management using a structured approach to goal-setting and outcome measurement: First cycle results from the ULIS-III Study. J Rehabil Med. 2021 Jan 1;53(1):jrm00133. doi: 10.2340/16501977-2770. PMID 33206198
- [Derived] Turner-Stokes L, Ashford S, Jacinto J, Maisonobe P, Balcaitiene J, Fheodoroff K. Impact of integrated upper limb spasticity management including botulinum toxin A on patient-centred goal attainment: rationale and protocol for an international prospective, longitudinal cohort study (ULIS-III). BMJ Open. 2016 Jun 17;6(6):e011157. doi: 10.1136/bmjopen-2016-011157. PMID 27315835